CLINICAL TRIAL: NCT01002547
Title: NAFLD in T2DM: Prevalence in Hispanics and Role of Treatment
Brief Title: Prevalence of Non-alcoholic Fatty Liver Disease (NAFLD) in Hispanics With Diabetes Mellitus Type 2 (T2DM) and Role of Treatment
Acronym: VA NASH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-015-08F; HSC20090401H (Other: IRB UTHSCSA); VA-ORD#GRANT00508571 (Other Grant/Funding Number: CSRD CSP); 610-2011 (Other: University of Florida IRB-01)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: steatohepatitis; type 2 diabetes; fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Placebo Comparator): Diabetic with proven NASH by biopsy
  Interventions: Drug: pioglitazone-placebo; Drug: Vitamin E-placebo
- Arm 2 (Active Comparator): Diabetic with proven NASH by biopsy
  Interventions: Drug: pioglitazone; Dietary Supplement: Vitamin E
- Arm 3 (Other): Diabetic with proven NASH by biopsy
  Interventions: Drug: pioglitazone-placebo; Dietary Supplement: Vitamin E

INTERVENTIONS:
Drug: pioglitazone-placebo — This is a RCT in which all patients will be educated on a -500 kcal/day diet and a healthy lifestyle. Depending on randomization, subjects adjudicated to placebo will be started at the same time as the active (pioglitazone) arm following completion of the baseline measurements and continued on placebo for the rest of the clinical trial.
  Arms: Arm 1
Drug: pioglitazone — Pioglitazone will be started on 30 mg/day, titrated to the maximal dose (45 mg/day) at two months and continued at this dose for the rest of the clinical trial.
  Other Names: Actos
  Arms: Arm 2
Dietary Supplement: Vitamin E — All participants will receive vitamin E 400 IU orally twice daily.
  Arms: Arm 2
Drug: pioglitazone-placebo — This is a RCT in which all patients will be educated on a -500 kcal/day diet and a healthy lifestyle. Depending on randomization, subjects adjudicated to placebo will be started at the same time as the active (pioglitazone) arm following completion of the baseline measurements and continued on placebo for the rest of the clinical trial.
  Arms: Arm 3
Dietary Supplement: Vitamin E — All participants will receive vitamin E 400 IU orally twice daily.
  Arms: Arm 3
Drug: Vitamin E-placebo — Placebo of vitamin E will be given to arm 3.
  Arms: Arm 1

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a chronic liver condition frequently associated with type 2 diabetes (T2DM) and characterized by insulin resistance and hepatic fat accumulation. Liver fat may range from simple steatosis to severe steatohepatitis with necroinflammation and variable degrees of fibrosis (nonalcoholic steatohepatitis or NASH). Up to 40% of patients with NAFLD develop NASH in recent series. Risk factors for progression to NASH are unclear, but appears to be more common and progress more rapidly in older individuals, and in the presence of obesity and T2DM. Because the VA population in San Antonio, Texas, frequently combine these risk factors for NASH it was felt that a study targeting this very high-risk population was needed.

This study will establish the long-term efficacy (primary endpoint: liver histology) and safety of pioglitazone for the treatment of VA patients with T2DM and NASH. All patients diagnosed with NASH will be offered lifestyle modification/weight loss (current standard of care) while being randomized to pioglitazone, vitamin E or placebo for up to 3 years. We believe that in such a high-risk population for complications from NASH, a substantial benefit may be expected from early detection and treatment.

Specifically, the arms are: a) pioglitazone + vitamin E; b) vitamin E + placebo of pioglitazone; c) placebo of both. Patients are randomized to one of these 3 arms, and followed in a double-blind fashion for up to 18 months. Patients are then offered to continue into an open-label phase with pioglitazone + vitamin E or vitamin E alone for another 18 months.

DETAILED DESCRIPTION:
Many NAFLD studies have found that the progression from "benign" steatosis to severe necroinflammation and cirrhosis as observed in NASH varies widely depending upon the initial stage at diagnosis, as well the presence or absence of specific risk factors associated with disease progression. The factors that promote necroinflammation and fibrosis development are complex, but are frequently associated with the presence of long-standing obesity, metabolic syndrome, and in particular, of T2DM. Indeed, hyperglycemia has been identified as the single most consistent factor for disease progression in many studies (Angulo et al, Hepatology 1999) Marceau et al, JCEM 1999; Luyckx et al, Obes Relat Metab Disord, 1998; Mofrad et al, Hepatology 2003; many others; reviewed by Cusi, Current Diabetes Reports, 2009).

Given the worse prognosis of NASH in patients with T2DM, it is quite surprising that few studies have focused on the prevalence of the disease and on early screening and treatment of patients with diabetes for NASH. A prospective study conducted by Gupte et al (Gastroenterology & Hepatology, 2004) reported biopsy-proven NASH in 87% of diabetics, 22% having moderate to severe disease. In a retrospective analysis of 44 patients with T2DM worked-up for NAFLD, Younussi et al also found that cirrhosis was more prevalent in diabetics vs. nondiabetics (25% vs. 10%, p<0.001) (Hepatology 2004). In recent years, the diagnosis of fatty liver has been made easier with the standardization of liver magnetic resonance and spectroscopy (MRS) which has allowed a fast and highly reproducible test for NAFLD. With this screening tool we have found that NAFLD is present in >80% of unselected patients with T2DM. In non-diabetic patients a handful of small studies with paired biopsies indicate that fibrosis progresses over time in 32-41% of patients with NAFLD (reviewed by Ali & Cusi, Annals of Medicine, 2009). Obesity and T2DM were the 2 most prominent factors of poor prognosis, while elevated liver enzymes (ALT or AST/ALT ratio) were of lesser value (Mofrad et al, Hepatology 2003; Sorrentino et al, Hepatology 2004; Kunde et al, Hepatology 2005).

This study aims at establishing the role of pioglitazone and of vitamin E in VA patients. Weight loss remains the standard of care because no therapy has conclusively proven to be effective in the long-term. Pharmacological therapies with modest effects have included pentoxifylline, orlistat, cytoprotective agents, ursodeoxycholic acid and lipid-lowering agents, while insulin-sensitizers such as metformin and thiazolidinediones have yielded more provocative results in small uncontrolled studies in NASH. Our research group recently demonstrated in a randomized, double-blind, placebo-controlled trial, that pioglitazone treatment for 6 months in patients with T2DM and NASH significantly improved glycemic control, glucose tolerance, insulin sensitivity and systemic inflammation (Belfort et al, NEJM 2006). This was associated with a ~50% decrease in steatohepatitis (p<0.001) and a 37% reduction of fibrosis within the pioglitazone-treated group (-37%, p<0.002), although this fell short of statistical significance when compared with placebo (p=0.08). Our results provided "proof-of-principle" that pioglitazone may be the first agent capable of altering the natural history of the disease. However, definitive proof requires establishing its safety and efficacy in a large number of subjects treated for a longer period of time. The CRN is conducting the PIVENS trial (www.ClinicalTrials.gov; NCT 00063622) examining the role of pioglitazone, vitamin E or placebo in NASH, but the study design excluded diabetics, only ~5% of patients were Hispanic and studied a younger population than that typical from VA Medical Centers. Also, this important multicenter trial did not perform the in-depth metabolic measurements this trial will carry out (i.e., insulin clamps with glucose turnover measurements, indirect calorimetry, etc.).

Understanding the long-term impact of thiazolidinediones and of vitamin E in patients with NASH and T2DM, who are believed to be at the highest risk for liver disease progression, will have important implications not only for the treatment of NASH but for drug selection and treatment algorithms in T2DM, as an insulin-sensitizer approach of pioglitazone (in addition to metformin) would be preferred over therapies such as sulfonylureas or insulin, if proven to be effective to treat NASH in T2DM. However, currently the most common strategy to treat T2DM is an insulin secretion-based approach (i.e., sulfonylureas and/or insulin) that has little impact on liver fat and promotes weight gain without a major improvement in insulin sensitivity, promoting chronic hyperinsulinemia and self-perpetuating the metabolic milieu that promotes hepatic lipogenesis and fatty liver disease. Therefore, understanding the role of pioglitazone and vitamin combined, of vitamin e alone (plus pioglitazone placebo tablets as control) and compared to a third arm with placebo of both (pioglitazone and vitamin E) is important to move the field forward.

Of note, the study started at the San Antonio VAMC, TX where ~60% of the population was Hispanic. However, once Dr. Kenneth Cusi (principal investigator) moved to the Gainesville VAMC, FL the study was transferred to Gainesville and recruitment continued in this new site where the prevalence of Hispanics is only 5% (75% Caucasians, 20% African American). Therefore, the final patient mix will reflect more the latter ethnic mix.

ELIGIBILITY:
Inclusion Criteria:

* Be able to communicate meaningfully with the Investigator and be legally competent to provide written informed consent.
* Subjects of both genders from within the Veterans Administration Healthcare System with an age range between 18 to 70 years (inclusive).
* Have type 2 diabetes mellitus as defined by the American Diabetes Association guidelines.
* Female volunteers must be non-lactating and must either be at least one year post-menopausal, or be using adequate mechanical contraceptive precautions (i.e. intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period.
* The following laboratory values:

  * Hemoglobin at least 12 gm/dl in males or 11 gm/dl in females, WBC count 3,000/mm3 (neutrophil count 1,500/mm3) and platelets 100,000/mm3
  * Albumin equal or greater than 3.0 g/dl
  * Serum creatinine less than 1.8 mg/dl
  * AST and ALT up to 3.0 times upper limit of normal and alkaline phosphatase 2.5 times ULN

Exclusion Criteria:

* Any cause of chronic liver disease other than NASH (such as -but not restricted to- alcohol or drug abuse, medication, chronic hepatitis B or C, autoimmune, hemochromatosis, Wilson's disease, alpha1-antitrypsin deficiency).
* Any clinical evidence or history of ascitis, bleeding varices, or spontaneous encephalopathy.
* History of alcohol abuse (alcohol consumption greater than 20 grams of ethanol per day) or a positive AUDIT screening questionnaire.
* Prior surgical procedures to include gastroplasty, jejunoileal or jejunocolic bypass.
* Prior exposure to organic solvents such as carbon tetrachloride.
* Total parenteral nutrition (TPN) within the past 6 months.
* Subjects with type 1 diabetes mellitus.
* Patients on chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for 4 weeks before entry into the study.
* Patients on drugs known to cause hepatic steatosis: estrogens or other hormonal replacement therapy, tamoxifen, raloxifene, oral glucocorticoids, chloroquine and others.
* Patients with a history of clinically significant heart disease (New York Heart Classification greater than grade II), peripheral vascular disease (history of claudication), or diagnosed pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation).
* Patients with severe osteoporosis (-3.0 at the level of spine and hip).
* Patients who have clinically significant acute or chronic medical conditions not specifically written in the protocol, but that based in the investigator's clinical judgment he/she considers unlikely that he will be able to complete study participation or that such participation may be potentially detrimental to his well-being.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-06-24 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cusi, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bril F, Biernacki DM, Kalavalapalli S, Lomonaco R, Subbarayan SK, Lai J, Tio F, Suman A, Orsak BK, Hecht J, Cusi K. Role of Vitamin E for Nonalcoholic Steatohepatitis in Patients With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2019 Aug;42(8):1481-1488. doi: 10.2337/dc19-0167. Epub 2019 May 21. PMID 31332029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the endocrinology and hepatology clinics at two VA Medical Centers (i.e., Audie L. Murphy in San Antonio, TX and Malcom Randall in Gainesville, FL). The study was conducted between June 2010 and September 2016 (recruitment was completed in December 2014).
Pre-assignment Details: After initial screening (medical history, physical exam, laboratories, 75-gram oral glucose tolerance test [OGTT]), patients were instructed to keep physical activity and diet constant during the run-in phase (mean duration: 1 month).
Groups:
- Placebo: Patients with T2DM and biopsy-proven NASH.
  Pioglitazone-placebo: This is a RCT in which all patients will be educated on a -500 kcal/day diet and a healthy lifestyle. Depending on randomization, subjects adjudicated to placebo will be started at the same time as the active (pioglitazone) arm and following the same up-titration. Placebo pills have the same characteristics as pills with active medication.
  Vitamin E-placebo: Placebo of vitamin E will be given to arm 1.
- Vitamin E: Patients with T2DM and biopsy-proven NASH.
  Pioglitazone-placebo: This is a RCT in which all patients will be educated on a -500 kcal/day diet and a healthy lifestyle. Depending on randomization, subjects adjudicated to placebo will be started at the same time as the active (pioglitazone) arm and following the same up-titration. Placebo pills have the same characteristics as pills with active medication.
  Vitamin E: All participants will receive vitamin E 400 IU orally twice daily.
- Pioglitazone + Vitamin E: Patients with T2DM and biopsy-proven NASH.
  Pioglitazone: This is a RCT in which all patients will be educated on a -500 kcal/day diet and a healthy lifestyle. Pioglitazone will be started on 30 mg/day, titrated to the maximal dose (45 mg/day) at two months and continued at this dose for the rest of the clinical trial.
  Vitamin E: All participants will receive vitamin E 400 IU orally twice daily.
Period: Overall Study
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Started | 32 | 36 | 37
Completed | 24 | 33 | 29
Not Completed | 8 | 3 | 8
Not completed — Withdrawal by Subject | 4 | 0 | 5
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Death | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E | Total
Number analyzed (Participants) | 32 | 36 | 37 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11) | 60 (9) | 60 (6) | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 7 | 12
  Male | 30 | 33 | 30 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 27 | 26 | 76
  African American | 2 | 4 | 3 | 9
  Hispanic | 7 | 5 | 8 | 20
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 33.6 (4.0) | 33.8 (4.6) | 35.2 (4.3) | 34.5 (4.2)
Total body fat [Mean (Standard Deviation); unit: percentage] | 36 (5) | 37 (6) | 38 (6) | 37 (6)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 153 (37) | 158 (41) | 144 (43) | 152 (44)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 7.2 (1.2) | 7.5 (1.3) | 7.3 (1.1) | 7.3 (1.2)
Use of glucose-lowering medications [Count of Participants; unit: Participants]
  Metformin | 27 | 29 | 29 | 85
  Sulfonylurea | 13 | 15 | 14 | 42
  Insulin | 8 | 10 | 10 | 28
Fasting plasma insulin [Mean (Standard Deviation); unit: uU/mL] | 18 (13) | 22 (14) | 16 (10) | 18 (13)
Fasting free fatty acids [Mean (Standard Deviation); unit: umol/ml] | 0.41 (0.15) | 0.39 (0.14) | 0.41 (0.15) | 0.40 (0.14)
Intrahepatic triglyceride content [Mean (Standard Deviation); unit: percentage] | 10.5 (5.8) | 11.7 (5.7) | 13.8 (8.4) | 12.2 (7.0)
Plasma AST [Mean (Standard Deviation); unit: U/L] | 40 (23) | 41 (22) | 32 (18) | 37 (21)
Plasma ALT [Mean (Standard Deviation); unit: U/L] | 53 (33) | 53 (32) | 40 (25) | 49 (31)
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 171 (40) | 174 (44) | 170 (53) | 172 (46)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dl] | 94 (33) | 98 (39) | 91 (44) | 94 (39)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dl] | 39 (10) | 39 (9) | 38 (10) | 38 (9)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dl] | 154 [117 to 255] | 156 [126 to 210] | 163 [108 to 274] | 158 [116 to 243]
Statin use [Count of Participants; unit: Participants] | 25 | 26 | 29 | 80
NAFLD activity score [Mean (Standard Deviation); unit: units on a scale] — Calculated as the sum of steatosis grade (0 to 3), inflammation grade (0 to 3), and ballooning grade (0 to 2). Therefore, this score ranges from 0 to 8.
  Steatosis: 0 = <5% fat; 1 = 5-33% fat; 2 = >33-66% fat; 3 = >66% fat.
  Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x.
  Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning.
  Fibrosis stage: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
  units on a scale | 4.2 (1.6) | 3.9 (1.6) | 3.7 (1.3) | 4.0 (1.5)
Steatosis [Mean (Standard Deviation); unit: units on a scale] — Steatosis range 0-3, where: 0 = <5% fat; 1 = 5-33% fat; 2 = >33-66% fat; 3 = >66% fat.
  units on a scale | 1.8 (0.7) | 1.7 (0.8) | 1.6 (0.8) | 1.7 (0.7)
Inflammation [Mean (Standard Deviation); unit: units on a scale] — Lobular Inflammation, range 0-3, where: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x.
  units on a scale | 1.6 (0.6) | 1.3 (0.5) | 1.4 (0.5) | 1.4 (0.6)
Hepatocyte ballooning [Mean (Standard Deviation); unit: units on a scale] — Hepatocyte Ballooning, range 0-2, where: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning.
  units on a scale | 0.9 (0.8) | 0.9 (0.8) | 0.7 (0.6) | 0.8 (0.7)
Fibrosis [Mean (Standard Deviation); unit: units on a scale] — Fibrosis stage, range 0-4, where: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
  units on a scale | 1.5 (1.0) | 1.6 (1.2) | 1.4 (1.1) | 1.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Liver Histology (Kleiner's et al Criteria, Hepatology 2005)
Description: Number of patients with reduction of at least 2 points in the nonalcoholic fatty liver disease activity score (NAS) (with reduction in at least 2 different histological categories) without worsening of fibrosis. NAS is the sum of the separate scores for steatosis (0-3), hepatocellular ballooning (0-2) and lobular inflammation (0-3), and ranges from 0-8 .
  The scoring system is based on the following grading:
  Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x. Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning. Fibrosis: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
Time Frame: 18 months
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 32 | 36 | 37
Participants | 7 | 13 | 24

2. Secondary Outcome: Number of Participants With Resolution of NASH Without Worsening of Fibrosis
Description: Resolution of NASH was defined as absence of NASH after 18 months of therapy in patients with definite NASH (presence of zone 3 accentuation of macrovesicular steatosis of any grade, hepatocellular ballooning of any degree, and lobular inflammatory infiltrates of any amount) at baseline.
Time Frame: Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 32 | 36 | 37
Participants | 5 | 14 | 20

3. Secondary Outcome: Mean Individual Histological Scores
Description: Mean change in individual scores compared to baseline. Steatosis range 0-3, where: 0 = <5% fat; 1 = 5-33% fat; 2 = >33-66% fat; 3 = >66% fat.
  Lobular Inflammation, range 0-3, where: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x.
  Hepatocyte Ballooning, range 0-2, where: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning.
  Fibrosis stage, range 0-4, where: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
Time Frame: Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 32 | 36 | 37
units on a scale
  Steatosis | -0.4 (0.9) | -1.0 (1.0) | -1.3 (1.0)
  Inflammation | -0.2 (0.8) | -0.4 (0.7) | -0.6 (0.7)
  Ballooning | -0.1 (0.9) | -0.5 (0.9) | -0.6 (0.9)
  Fibrosis | -0.3 (1.1) | -0.6 (1.0) | -0.6 (0.9)

4. Secondary Outcome: Individual Histological Scores
Description: Number of patients with improvement of at least 1 grade in each of the histological parameters.
  Steatosis: 0 = <5%; 1 = 5-33%; 2 = >33-66%; 3 = >66%. Lobular Inflammation: 0 = No foci 1 = <2 foci/200x; 2 = 2-4 foci/200x, 3 = >4 foci/200x.
  Hepatocyte Ballooning: 0 = None; 1 = Few balloon cells; 2 = Many cells/prominent ballooning.
  Fibrosis: 0 = None; 1 = Perisinusoidal or periportal; 2 = Perisinusoidal and portal/periportal; 3 = Bridging fibrosis, 4 = Cirrhosis.
Time Frame: Month 18
Population: Multiple imputation was used to impute missing histologic data for patients who did not complete 18 months of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 32 | 36 | 37
Participants
  Steatosis | 15 | 24 | 32
  Inflammation | 14 | 13 | 25
  Ballooning | 11 | 18 | 23
  Fibrosis | 10 | 19 | 19

5. Secondary Outcome: Liver Fat by Magnetic Resonance Imaging and Spectroscopy (MRS).
Description: Change from baseline in intrahepatic triglyceride content after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of therapy
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
percentage | 1 (7) | -6 (6) | -10 (6)

6. Secondary Outcome: Weight
Description: Change from baseline in weight
Time Frame: Month 18
Population: Patients completing 18 months of follow-up
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
kg | -0.8 (4.2) | 0.5 (5.6) | 5.7 (5.4)

7. Secondary Outcome: Body Mass Index
Description: Weight (in kg) / (Height [in m] x Height [in m])
Time Frame: Month 18
Population: Patients completing 18 months of follow-up.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
kg/m2 | -0.6 (1.6) | 0.1 (2.3) | 1.4 (1.6)

8. Secondary Outcome: Total Body Fat by DEXA
Description: Change from baseline in total body fat by DEX after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of follow-up
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
percentage | 0 (3) | 0 (3) | 2 (3)

9. Secondary Outcome: Plasma AST
Description: Change from baseline in plasma AST after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of follow-up
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
U/L | -8 (28) | -15 (20) | -10 (10)

10. Secondary Outcome: Plasma ALT
Description: Change from baseline in plasma ALT after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of follow-up
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
U/L | -6 (42) | -24 (29) | -18 (17)

11. Secondary Outcome: Fasting Plasma Glucose
Description: Change from baseline after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of therapy
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
mg/dl | 6 (53) | -3 (39) | -16 (36)

12. Secondary Outcome: Fasting Plasma Insulin
Description: Change from baseline after 18 months of therapy
Time Frame: Month 18
Population: Patients completing 18 months of follow-up, not on insulin therapy
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 16 | 18 | 19
uU/ml | 3 (12) | -3 (6) | -3 (6)

13. Secondary Outcome: Matsuda Index
Description: This is a method for assessing insulin resistance (IR) based on measurements of glucose and insulin during the oral glucose tolerance test. The formula used is = (10000/(SQRT(fasting plasma glucose * fasting plasma insulin * ((fasting plasma glucose * 15 + glucose at minute 30 * 30 + glucose at minute 60 * 30 + glucose at minute 90 * 30 + glucose at minute 120 * 15)/120)*((fasting plasma insulin * 15 + insulin at minute 30 * 30 + insulin at minute 60 * 30 + insulin at minute 90 * 30 + insulin at minute 120 * 15)/120))), with a lower value representing worse insulin resistance.
Time Frame: Month 18
Population: Patients completing 18 months of follow-up, not on insulin therapy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 16 | 18 | 19
units on a scale | 2.53 (0.39) | 2.31 (0.29) | 4.02 (0.72)

14. Secondary Outcome: Total Cholesterol
Description: Change from baseline in plasma total cholesterol after 18 months of therapy
Time Frame: Month 18
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
mg/dl | -11 (31) | 5 (29) | 1 (43)

15. Secondary Outcome: Triglycerides
Description: Change from baseline in plasma triglycerides after 18 months of therapy
Time Frame: Month 18
Population: All patients completing 18 months of follow-up
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
mg/dl | 13 [-2 to 46] | 14 [-28 to 74] | -2 [-48 to 31]

16. Secondary Outcome: HDL-cholesterol
Description: Change from baseline in plasma HDL-cholesterol after 18 months of therapy
Time Frame: Month 18
Population: All patients completing 18 months of follow-up
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
mg/dl | -1 (4) | 1 (4) | 3 (7)

17. Secondary Outcome: LDL-cholesterol
Description: Change from baseline in plasma LDL-cholesterol after 18 months of therapy
Time Frame: Month 18
Population: All patients completing 18 months of therapy
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
Number analyzed (Participants) | 24 | 33 | 29
mg/dl | -12 (31) | 0 (30) | -4 (31)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the entire period of the randomized controlled trial (18 months).
Description: Specific questionnaire focused on weight changes, peripheral edema, fractures, and GI disturbances.
Arm/Group | Placebo | Vitamin E | Pioglitazone + Vitamin E
All-Cause Mortality (participants affected / at risk) | 0/32 | 2/36 | 2/37
Serious Adverse Events (participants affected / at risk) | 5/32 | 6/36 | 12/37
Other Adverse Events (participants affected / at risk) | 15/32 | 18/36 | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Vitamin E (N=36) | Pioglitazone + Vitamin E (N=37)
Arrhythmia (Cardiac disorders) | 1 | 1 | 1
Hypertensive crisis (Cardiac disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1
Hypertriglyceridemia (Endocrine disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar abscess (Infections and infestations) | 0 | 0 | 1
Endocarditis (Cardiac disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Subdural hematoma (Nervous system disorders) | 0 | 1 | 0
Biopsy-related complications (Gastrointestinal disorders) | 2 | 1 | 2
Back, joint, or hernia repair surgery (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Diagnosis of prostate cancer (Renal and urinary disorders) | 0 | 0 | 1
Asthma/COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Vitamin E (N=36) | Pioglitazone + Vitamin E (N=37)
Atypical chest pain or epigastralgia (Cardiac disorders) | 3 | 4 | 6
Lower limb edema (Cardiac disorders) | 1 | 0 | 5
Diarrhea/constipation (Gastrointestinal disorders) | 6 | 6 | 4
AST/ALT elevations (Hepatobiliary disorders) | 3 | 1 | 0
Upper respiratory infection, sinusitis, bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3
Unspecific dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 7
Hypoglycemia (Endocrine disorders) | 6 | 7 | 13
Bone fractures (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Back or joint pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 9

LIMITATIONS AND CAVEATS:
Relative small sample size. A larger sample size could have resulted in significantly positive results for vitamin E alone in secondary outcomes. Because of this we acknowledge that vitamin E may still be an alternative for some patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No